CLINICAL TRIAL: NCT04396808
Title: Genomics in Michigan to AdJust Outcomes in Prostate canceR (G-MAJOR): A Randomized Multi-center Study for Men With Newly Diagnosed Favorable Risk Prostate Cancer
Brief Title: Genomics in Michigan to AdJust Outcomes in Prostate canceR (G-MAJOR) for Men With Newly Diagnosed Favorable Risk Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Myrexis Inc. (Industry); Veracyte, Inc. (Industry); MDx Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UMCC 2019.132; HUM00173277 (Other: University of Michigan)
Record Dates: First submitted 2020-05-15; First posted 2020-05-21 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Biomarkers; Active surveillance; Gene Expression Classifier
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: 1:1 cluster-crossover in 3 month blocks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of care (no pre-treatment genomics testing) (Active Comparator): Provider will discuss askMUSIC results with patient prior to deciding on a management strategy (standard of care).
  Interventions: Other: Standard of care (askMUSIC score)
- Standard of care + pre-treatment genomics testing (Active Comparator): Provider will discuss askMUSIC and Gene Expression Classifier (GEC) results with patient prior to deciding on a cancer management strategy. Patients' biopsy tissue will be analyzed using one of the following GECs: Decipher, Prolaris or Oncotype Dx.
  Interventions: Device: Decipher; Device: Prolaris; Device: Oncotype Dx Genomic Prostate Score (GPS); Other: Standard of care (askMUSIC score)

INTERVENTIONS:
Device: Decipher — The Decipher test (GenomeDx Biosciences) is a genomic test that will be performed on prostate biopsy tissue. Results will be provided to the patient and physician prior to making a treatment decision.
  Other Names: Decipher Prostate Cancer Classifier
  Arms: Standard of care + pre-treatment genomics testing
Device: Prolaris — The Prolaris test (Myriad Genetics, Inc.) is a genomic test that will be performed on prostate biopsy tissue. Results will be provided to the patient and physician prior to making a treatment decision.
  Other Names: Prolaris Prostate Cancer Test
  Arms: Standard of care + pre-treatment genomics testing
Device: Oncotype Dx Genomic Prostate Score (GPS) — The Oncotype Dx GPS test (Exact Sciences corp.) is a genomic test that will be performed on prostate biopsy tissue. Results will be provided to the patient and physician prior to making a treatment decision.
  Arms: Standard of care + pre-treatment genomics testing
Other: Standard of care (askMUSIC score) — AskMUSIC is a risk calculator based on standard clinical and pathologic variables (https://ask.musicurology.com/) and is generally included as part of routine clinical care.
  Other Names: askMUSIC score

SUMMARY:
This study seeks to determine the clinical impact of Gene Expression Classifier (GEC) testing in prostate cancer care while also developing a pragmatic approach for improved GEC clinical use and future study.

DETAILED DESCRIPTION:
All patients in this study have received or will receive a score from the Michigan Urological Surgery Improvement Collaborative's Cancer of the Prostate Risk Assessment (askMUSIC) scoring system, at the time of enrollment. AskMUSIC is a risk calculator based on standard clinical and pathologic variables and is generally included as part of routine clinical care. The variables used in the risk calculator are prostate-specific antigen (PSA), Gleason score, number of positive core biopsies, number of negative core biopsies, and clinical stage.

Patients will be randomized to either an intervention arm or a control arm. In the control arm, the treating provider will review the askMUSIC score with the patient. In the intervention arm, the treating provider will review the askMUSIC and the GEC score with the patient. Biopsies obtained during the course of standard clinical care will be analyzed using one of the following GECs: Decipher, Prolaris or Oncotype Dx Genomic Prostate Score. No additional biopsies will be obtained as part of this study.

After reviewing the results, patients and their treating physicians will decide on a management strategy.

Long-term follow-up will be tracked through the Michigan Urological Surgery Improvement Collaborative (MUSIC) registry.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients who have undergone diagnostic prostate biopsy in the past 9 months.
* Prostate biopsy tumor tissue (FFPR block) available for processing
* Age 18 years or older
* PSA <20 ng/ml
* Grade Group (GG) 1 cancer with > 2 biopsy cores involved with cancer OR GG2 cancer
* Ability to understand and the willingness to sign a written informed consent. A subject's legally acceptable representative may sign the consent form.

Exclusion Criteria:

* Clinical (on digital rectal exam) or radiographic evidence (if MRI performed) of T3 disease
* Nodal or metastatic prostate cancer (if staging imaging performed)
* Prior prostate cancer treatment, including prostatectomy, radiation therapy, or hormone therapy.
* Prior prostate gene expression classier testing

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2031-04-30 (Estimated)

PRIMARY OUTCOMES:
Binomial proportion of men on active surveillance without treatment | At 2 years

SECONDARY OUTCOMES:
Occurence of grade reclassification | At 2 years
  Grade reclassification defined as an increase in grade group on surveillance biopsy (GG=1 to GG≥2 or GG=2 to GG≥3) for patients managed on active surveillance
Rate of indolent pathology | At time of prostatectomy (for patients who undergo procedure), up to 2 years
  To determine the impact of GEC testing on the rate of potentially unnecessary surgery, as defined by indolent pathology at prostatectomy (GG1 and stage pT2).
Mean score per arm of patient reported urinary function questionnaire | At 2 years
  Assessed by patient reported Expanded Prostate Cancer Index (EPIC) Urinary Incontinence Domain (UIN) questionnaire. Response options form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better quality of life (QOL).
Proportion of patients with changes from baseline in urinary function exceeding Minimal Important Differences (MID). | Baseline to 12 months and 2 years
  Assessed by patient reported EPIC UIN questionnaire. For this measure, MID = 9 points.
Mean score per arm of patient reported sexual function questionnaire | At 2 years
  Assessed by patient reported Expanded Prostate Cancer Index (EPIC) sexual domain questionnaire. Response options form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better QOL.
Proportion of patients with changes from baseline in sexual function exceeding Minimal Important Differences (MID). | Baseline to 12 months and 2 years
  Assessed by patient reported EPIC sexual function questionnaire. For this measure, MID = 11 points.
Time to biochemical recurrence (BCR) | From time of radical therapy until the event or the last measured follow-up, up to 2 years
  Time from treatment PSA >= 0.2 ng/mL for patients undergoing surgery (with PSA at least 5 weeks after surgery) and nadir plus 2.0 ng/mL for patients undergoing radiotherapy.
Time to distant metastases | From time of radical therapy until the event or the last measured follow-up, up to 2 years
  Assessed by CT, MRI, bone scan, and/or PET scan
Mean score per arm of health-related quality of life (HRQOL) | At 2 years
  Assessed by patient reported Expanded Prostate Cancer Index Composite short form (EPIC-26). EPIC-26 encompasses 5 domains (Urinary Incontinence, Urinary Irritative/Obstructive, Bowel, Sexual, and Hormonal). Response options for each of 26 items form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better HRQOL.
Rate of adverse pathology at prostatectomy | At time of prostatectomy, up to 5 years from enrollment
  To determine the performance of GEC testing in predicting adverse pathology, defined as GG≥3 and/or ≥pT3 disease.
Rate of biochemical recurrence | Up to 5 years following treatment
  To determine the performance of GEC testing in predicting biochemical recurrence, defined as PSA >= 0.2 ng/mL for patients undergoing surgery (with PSA at least 5 weeks after surgery) and nadir plus 2.0 ng/mL for patients undergoing radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Morgan, M.D., Principal Investigator — University of Michigan; Daniel Spratt, M.D., Principal Investigator — University of Michigan
Locations (8):
- United States (8):
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Sherwood Medical Center, Detroit, Michigan
  - Spectrum Health Medical Group, Grand Rapids, Michigan
  - Western Michigan Urological Associates, Holland, Michigan
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vince RA Jr, Jiang R, Qi J, Tosoian JJ, Takele R, Feng FY, Linsell S, Johnson A, Shetty S, Hurley P, Miller DC, George A, Ghani K, Sun F, Seymore M, Dess RT, Jackson WC, Schipper M, Spratt DE, Morgan TM. Impact of Decipher Biopsy testing on clinical outcomes in localized prostate cancer in a prospective statewide collaborative. Prostate Cancer Prostatic Dis. 2022 Apr;25(4):677-683. doi: 10.1038/s41391-021-00428-y. Epub 2021 Jul 20. PMID 34285350